CLINICAL TRIAL: NCT00255502
Title: A Safety, Tolerability and Pharmacokinetics Study of TOPROL-XL® (Metoprolol Succinate) Extended-release Tablets (Metoprolol CR/XL) in Hypertensive Pediatric Subjects: A Multicenter, Open-Label Extension of Protocol 307A
Brief Title: 307B - Safety, Tolerability and Pharmacokinetics Study of TOPROL-XL® in Hypertensive Pediatric Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4020C00001; 307B
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2006-11

CONDITIONS: Hypertension
Keywords: Pediatric hypertension
MeSH Terms: conditions — Hypertension | interventions — Metoprolol

INTERVENTIONS:
Drug: metoprolol succinate

SUMMARY:
This was a 52-week, multicenter, open-label study to determine the safety, tolerability and pharmacokinetics of TOPROL-XL (metoprolol succinate) extended-release tablets (metoprolol CR/XL) in hypertensive pediatric subjects. The study population included school age children (age 6 to 12 years < Tanner Stage 3) and adolescents (> 12 years old or > Tanner Stage 3 to 16 years old) of both genders. Because response to some therapies in adult hypertension appears to be different in black and non-black populations, the recruitment will have a mixture of black and non-black subjects. Pharmacokinetic measurements were performed on a subset of patients. Thirty subjects (15 subjects each in the 6 to 12 year age group and the 13 to 16 year age group) had a series of blood samples drawn. All subjects had a trough plasma level taken 24 hours after the last dose of open-label metoprolol CR/XL (Visit 18) with the exception of those subjects who completed Protocol 307B (16 week open-label treatment).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 6 and 16 years inclusive at the time of screening.
* Have a negative urine pregnancy test, if female of childbearing potential. Have a signed informed consent by a parent or a legal guardian and an assent form signed by the subject (if applicable).
* Have hypertension that is either:

  1. Have successfully completed Protocol 307A, or, or
  2. Have dropped out of Protocol 307A or failed screening for Protocol 307A for sitting SBP/DBP greater than 20/10 mm Hg over the 95 th percentile using height adjusted charts for age and gender (see Appendices B through E inclusive), or
  3. Have not enrolled in Protocol 307A but meet all screening criteria for Protocol 307B and are enrolled at sites that have already randomized 6 subjects into Protocol 307A.
* Have the ability to swallow tablets.

Exclusion Criteria:

* Have secondary hypertension due to coarctation of aorta, pheochromocytoma, hyperthyroidism or Cushing's syndrome.
* Have a heart rate < 55 beats per minute at Visit 1.
* Have a history of asthma and/or recurring pulmonary disease or infections.
* Have a history of cystic fibrosis.
* Have a known hypersensitivity reaction to beta-blockers.
* Have a known bleeding, coagulation or platelet disorder that can interfere with blood sampling.
* Have a history of Insulin Dependent Diabetes Mellitus.
* Be in any situation or have any condition which, in the opinion of the investigator or sponsor, may interfere with participation in the study or produce a significant risk to the subject or interfere with the assessment of safety and efficacy endpoints.
* Have received any investigational agent for any therapeutic reason within 30 days prior to receiving study medication.
* Have a clinically significant cardiac valvular disease.
* Have a diagnosis of heart failure.
* Have clinically significant arrhythmia. This is defined as any arrhythmia requiring medical therapy or that causes symptoms.
* Atrioventricular (AV) conduction disturbance, ie, second or third degree AV block.
* Be unable or unwilling to comply with the study requirements.
* Be non-compliant during the single-blind placebo run-in period of the study as defined by missing three or more doses between study visits.
* Have impaired liver function defined as either acute liver disease or chronic liver disease with persistent liver enzyme values greater than one and one half times the upper limit of the normal range for AST or ALT.
* Have a known history of bilateral renal artery stenosis, or unilateral renal artery stenosis to a single kidney. Nephrotic subjects who are not in remission should be excluded.
* Be pregnant or breast-feeding an infant.
* Currently taking medications known to inhibit CYP2D6, such as quinidine, fluoxetine, paroxetine and propafenone.
* Currently taking catecholamine-depleting medications such as reserpine. For any subject who is currently taking medications known to inhibit CYP2D6 or any catecholamine-depleting medication, the sponsor must be contacted to assess feasibility for inclusion into the study.
* Currently taking any selective serotonin re-uptake inhibitors (SSRIs) or atypical antipsychotic medication.
* Have a history of alcohol or drug abuse, or have a positive urine screen for drugs of abuse or alcohol.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2002-07

PRIMARY OUTCOMES:
The purpose of this trial is to evaluate the pharmacokinetics and long term safety and
tolerability of metoprolol CR/XL in hypertensive pediatric subjects.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Toprol Medical Science Director, MD, Study Director — AstraZeneca
Locations (31):
- United States (30):
  - Research Site, Little Rock, Arkansas
  - Research Site, Bellflower, California
  - Research Site, Beverly Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Hartford, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Livingston, New Jersey
  - Research Site, New Hyde Park, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Beaumont, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
- Research Site, Santa Domingo, Dominican Republic

REFERENCES:
- [Derived] Batisky DL, Sorof JM, Sugg J, Llewellyn M, Klibaner M, Hainer JW, Portman RJ, Falkner B; Toprol-XL Pediatric Hypertension Investigators. Efficacy and safety of extended release metoprolol succinate in hypertensive children 6 to 16 years of age: a clinical trial experience. J Pediatr. 2007 Feb;150(2):134-9, 139.e1. doi: 10.1016/j.jpeds.2006.09.034. PMID 17236889